CLINICAL TRIAL: NCT06038864
Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema: Development of an Evaluation Set for Patients With LLL
Brief Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema: Aim 4
Acronym: EvaLymph-Leg4
Status: Recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Nij Smellinghe Hospital Drachten (Unknown)
Responsible Party: Principal Investigator, Tessa De Vrieze, Principal investigator, KU Leuven
Other Study IDs: s66033-aim4
Record Dates: First submitted 2023-09-04; First posted 2023-09-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lower Limb Lymphedema
Keywords: lymphedema; measurement; clinical evaluation
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive group: Patients with lower limb lymphoedema planned for intensive treatment
  Interventions: Diagnostic Test: 2 clinical evaluations with 1 month in between
- Maintenance group: Patients with stable lower limb lymphoedema who are in the maintenance phase (at least 3 months)
  Interventions: Diagnostic Test: 2 clinical evaluations with 1 month in between

INTERVENTIONS:
Diagnostic Test: 2 clinical evaluations with 1 month in between — Patients will be evaluated twice with all evaluation methods selected by the international expert group (cfr. aim 1) showing sufficient reliability and feasibility in the patient group with LLL from aim 1

SUMMARY:
Research investigating measurement properties for evaluating the decongestive treatment effect on different edema characteristics (e.g. water volume, hardness of the skin, water content,..) at the level of the lower limbs is missing. Information about the clinical relevant change criteria after treatment for nearly all these edema characteristics, is not present and requires investigation.

To assess the merits of each treatment in a reproducible manner, a reliable way of measuring limb volume and other edema characteristics must be established, as the evaluation of treatment effects without appropriate tools might lead to biased treatment effects.

First of all, in clinical practice, it is of utmost importance to know which edema characteristics need to be evaluated in order to assess the clinical evolution of a patient with lymphedema during and after treatment. Secondly, in order to draw proper conclusions about the treatment effect, it is necessary that to know from which criterion (or cut-off value) one can speak of a real clinical change for a certain lymphedema characteristic. Given that the edema characteristics that are most responsive to treatment and their corresponding criteria for clinically significant and relevant changes at the lower limbs have never been investigated before, the need for this research is high.

Therefore, the research questions in this study are: Which measurement tool(s) are able to detect clinically relevant changes in the lymphedema characteristics after the intensive treatment and during the maintenance treatment? When can a clinician speak of a clinically relevant change?

ELIGIBILITY:
Inclusion Criteria:

* Intensive treatment group

  * Unilateral or bilateral, primary or secondary LLL
  * No active metastases
  * If cancer-related lymphedema, time interval since surgery/ radiotherapy/ chemotherapy is ≥3 months
  * Objective diagnosis of lymphedema: ≥ 5% volume difference OR ≥ 2 minor/ 1 major criteria on lymphoscintigraphy OR presence of ICG dermal backflow
  * Age ≥ 18 years
  * Able to read, understand and speak Dutch
  * Planned to start with intensive decongestive lymphatic therapy at one or both legs
* Maintenance treatment group

  * See inclusion criteria 'intensive treatment group'
  * But: instead of patients planned to start with intensive lymphatic therapy, patients of this group should have ended their intensive treatment phase at least 3 months ago (= currently receiving maintenance decongestive lymphatic therapy)

Exclusion Criteria:

* Pregnant participants
* Presence of chronic venous insufficiency C4, C5, C6; deep venous thrombosis; post-thrombotic syndrome
* Presence of skin infections of wounds at the level of the lower limbs at the moment of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive treatment group: Patients planned to start with intensive decongestive lymphatic therapy at one or both legs.
  Maintenance treatment group: patienst who have ended their intensive treatment phase at least 3 months ago (= currently receiving maintenance decongestive lymphatic therapy)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of measurement methods | 1 month
  Sensitivity of measurement methods (resulting from aim 1:NCT05269264) in the evaluation of the treatment effect over time in patients with unilateral and bilateral LLL.
  Patients will be evaluated twice with 1 month in between.
Specificity of measurement methods | 1 month
  Specificity of measurement methods (resulting from aim 1:NCT05269264) in the evaluation of the treatment effect over time in patients with unilateral and bilateral LLL.
  Patients will be evaluated twice with 1 month in between.
Diagnostic accuracy of measurement methods | 1 month
  Diagnostic accuracy (in terms of area under the curve using a ROC curve, as well as sensitivity and specificity) of measurement methods (resulting from aim 1:NCT05269264) in the evaluation of the treatment effect over time in patients with unilateral and bilateral LLL.
  Patients will be evaluated twice with 1 month in between.

SECONDARY OUTCOMES:
Lymphedema volume after 4 weeks of intensive DLT in patients with unilateral and bilateral LLL | 1 month
  Evaluation of different outcome parameters in the patients from the 'intensive group' with unilateral LLL and patients with bilateral LLL:
  Lymphedema volume (foot, leg)
Hardness of skin after 4 weeks of intensive DLT in patients with unilateral and bilateral LLL | 1 month
  Evaluation of different outcome parameters in the patients from the 'intensive group' with unilateral LLL and patients with bilateral LLL:
  skin hardness test at the level of the foot, leg and midline region. Skin is palpated with thumb and index (and, if possible, compared to the contralateral side) Outcome: If skin is hardened; yes(1), otherwise; no(0)
Piiting status after 4 weeks f intensive DLT in patients with unilateral and bilateral LLL | 1 month
  Evaluation of different outcome parameters in the patients from the 'intensive group' with unilateral LLL and patients with bilateral LLL:
  Pitting test at the level of the foot, leg and midline region;
  The grading of edema is determined by pit depth (measured visually) and recovery time from grade 0-3. The scale is used to rate the severity and the scores are as follows:
  - Grade 0: No clinical edema- Grade 1: Slight pitting (up to 2 mm depth) - Grade 2: Moderate pitting (2-5 mm) - Grade 3: Noticeably deep pit (>5 mm)
Skinfold thickness after 4 weeks of intensive DLT in patients with unilateral and bilateral LLL | 1 month
  Evaluation of different outcome parameters in the patients from the 'intensive group' with unilateral LLL and patients with bilateral LLL:
  Skinfold test at the level of the foot, leg and midline region:
  Skin and subcutaneous tissue is lifted between thumb and index(and, if possible, compared to the contralateral side) Outcome:If skinfold is increased; yes(1), otherwise; no(0)
Extracellullar fluid after 4 weeks of intensive DLT in patients with unilateral and bilateral LLL | 1 month
  Evaluation of different outcome parameters (ECW ratio, total body water, body water left/right leg, ICW total/left/right, ECW total/left/right, phase angle total/left/right, impedance at 5 kHz) in the patients from the 'intensive group' with unilateral LLL and patients with bilateral LLL:
  Extracellular fluid
Problems in functioning after 4 weeks of intensive DLT in patients with unilateral and bilateral LLL | 1 month
  Disease-specific QoL (i.e. problems in functioning will be evaluated with the Lymph-ICF-LL.
  The Lymph-ICF-LL is a descriptive, evaluative tool containing 28 questions about impairments in function, activity limitations, and participation restrictions in patients with lower limb lymphedema. The questionnaire has 5 domains: physical function, mental function, general tasks/household activities, mobility activities, and life domains/social life.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa De Vrieze, Dr., Principal Investigator — KU Leuven
Locations (2):
- University Hospitals of Leuven, Leuven, Belgium
- Nij Smellinghe Hospital, Drachten, Netherlands